CLINICAL TRIAL: NCT07280585
Title: STOP-PKD: SGLT2-inhibition to Improve Prognosis in Polycystic Kidney Disease
Acronym: STOP-PKD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cologne (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Roman Müller, Prof. Dr. med., University Hospital of Cologne
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Uni-Koeln-5522; 2025-521276-59-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-24; First posted 2025-12-12 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Polycystic Kidney, Autosomal Dominant
Keywords: STOP-PKD; ADPKD; Dapagliflozin; SGLT2; PKD; polycystic kidney disease; SGLT2i; sodium-glucose; sodium glucose; Phase 3
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Polycystic Kidney Diseases | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Phase III, investigator-driven, multi-center, randomized, placebo-controlled, double-blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin 10 mg (Experimental)
  Interventions: Drug: Dapagliflozin 10 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: Dapagliflozin 10 mg — Participants receive 10 mg of Dapagliflozin orally once daily for 36 months.
  Arms: Dapagliflozin 10 mg
Drug: Matching Placebo — Participants receive a matching placebo orally once daily for 36 months.
  Arms: Placebo

SUMMARY:
Autosomal dominant polycystic kidney disease is the most common genetic cause of kidney failure. The only approved treatment for ADPKD - tolvaptan - is limited in its use by massive therapy-associated polyuria. This trial tests if the SGLT2-inhibitor dapagliflozin slows down the loss of kidney function in ADPKD.

DETAILED DESCRIPTION:
ADPKD is a genetic disease characterized by the growth of fluid-filled renal cysts, leading to progressive loss of kidney function. SGLT2- inhibitors have recently become available for the treatment of chronic kidney disease (CKD). The landmark trials, which proved the positive effect of SGLT2-inhibitors in CKD, excluded patients with ADPKD. Accordingly, current ADPKD-guidelines do not recommend the use of SGLT2-inhibitors in ADPKD.

This investigator-driven, randomized, placebo-controlled, multi-center, double-blind trial will assess the effect of daily dapagliflozin (10mg) intake on the chronic eGFR-slope in 420 patients with ADPKD. As a secondary endpoint the study will assess a composite endpoint triggered by reaching either 40%-eGFR loss, kidney failure or renal death. Safety aspects will additionally be addressed by an interim safety analysis considering total kidney volume, eGFR and copeptin-levels.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with ADPKD (modified Ravine criteria) ≥ 18 and ≤ 60 years
* Patients 18 - 39 years: eGFR ≥25 ml/min; patients 40 - 60 years: eGFR ≥25 and <90 ml/min/1.73 m2
* Indicators of rapid progression, either of the following:
* Mayo class 1D-E
* Mayo class 1C AND EITHER

  1. Truncating PKD1 mutation OR
  2. eGFR loss > 3ml/min/year (determined by ≥ 4 creatinine values within 4 years, ≥ 6 months measurement intervals) OR
  3. PROPKD score > 6 (patient history)
* IF patient is on ACE-I /ARBs: stable dose for 4 weeks before screening

Exclusion Criteria:

* Treatment with tolvaptan, somatostatin analogue, lithium or SGLT2i within the last 3 months before screening
* Medical history of diabetic ketoacidosis, necrotizing fasciitis or organ transplantation
* Diabetes mellitus type 1 or any type of diabetes mellitus due to insulin deficiency
* Uncontrolled ongoing urinary tract or genital infections
* Known intolerance of the study medication ingredients
* Uncontrolled grade 2 hypertension (>160/100 mmHg)
* Symptomatic hypotension, or systolic blood pressure <90 mmHg
* Primary renal disease other than ADPKD
* Hepatic impairment (aspartate transaminase [AST] or alanine transaminase [ALT]>3x the up-per limit of normal [ULN]; or total bilirubin >2x ULN at time of enrolment)
* Pregnancy, breastfeeding or women of child-bearing potential not using effective contraception method
* Not able to comply with the study protocol, in the investigator's judgement
* Not able to provide informed consent
* Participation in any other interventional clinical trial in the last 2 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 420 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2030-05-15 (Estimated); Study Completion 2030-05-15 (Estimated)

PRIMARY OUTCOMES:
Chronic eGFR slope | week 6 up to week 156 (end of treatment)
  The annual chronic eGFR slope will be calculated using all available serum creatinine values from week 6 to week 156 (end of treatment), using linear mixed models.

SECONDARY OUTCOMES:
Change in eGFR from pre-treatment to post-treatment (off-treatment values) | Week -4 to Week 168
  Change in kidney function will be assessed by comparing the mean eGFR values before treatment (calculated as the average of serum creatinine measurements at week -4 and week 0) with the mean eGFR values after treatment (calculated as the average of measurements at week 162 and week 168). The difference between these two timepoints represents the off-treatment change in kidney function.
Time to first occurrence of a composite renal endpoint | From randomization (week 0) until end of follow-up (up to week 168)
  Time from randomization to the first occurrence of any of the following events:
  1. A sustained ≥40% decrease in eGFR from randomization, confirmed by a second measurement at the next scheduled visit or measured at the last scheduled visit before death or study end.
  2. End-stage kidney disease (ESKD), defined as initiation of chronic dialysis, kidney transplantation, or a sustained eGFR <15 mL/min/1.73 m².
  3. Renal death.
Incidence of serious adverse events (SAEs) | From randomization (week 0) until end of follow-up (week 168)
  All serious adverse events (SAEs) will be collected.
Incidence of adverse events of special interest (AESIs) | From randomization (week 0) until end of follow-up (week 168)
  All adverse events of special interest (AESIs) will be collected.
Change in total kidney volume (TKV) after 1 year | Baseline (week -4 until week 0) to week 48 (first 150 patients)
  In the first 150 enrolled participants, total kidney volume (TKV) will be measured at baseline and at week 48 using standardized MRI protocols. The change in TKV over 48 weeks will be used to assess potential effects of dapagliflozin on kidney size.

OTHER OUTCOMES:
Change in kidney function based on cystatin-C measurements | week -4 until EOS (week 168)
  Annual slopes of eGFR decline (in mL/min/1,73m2 per year), as calculated with linear mixed models using all available cystatin-c values:
  1. on-treatment between week 6 and EOT (week 156)
  2. off-treatment: before treatment (week -4 and week 0) and after treatment (week 162 and week 168)
  3. between baseline and EOT (week 0-156)
Changes in albuminuria | from randomization (week 0) until EOT (week 156)
  Worsening (increase >50% in comparison to baseline) or new onset of albuminuria (defined as >30mg albumin/g creatinine)
Incidence of kidney stones | from randomization (week 0) until EOS (week 168)
  Number of symptomatic kidney stones (number of symptomatic episodes)
Total eGFR slope | from randomization (week 0) until week 156
  Total slope: annual slope of eGFR decline (in mL/min/1,73m2 per year), as calculated with linear mixed models, using all available creatinine values from baseline until end of treatment (week 0-156)

CONTACTS AND LOCATIONS:
Locations (27):
- Austria (2):
  - Vorarlberger Krankenhaus-Betriebsgesellschaft, Feldkirch
  - Medizinische Universitaet Innsbruck, Innsbruck
- Germany (20):
  - Universitaetsklinikum Aachen AöR, Aachen
  - Charite Universitaetsmedizin Berlin KöR, Berlin
  - Universitätsklinikum Köln, Cologne
  - Klinikum Dortmund gGmbH, Dortmund
  - Universitaetsklinikum Carl Gustav Carus Dresden an der Technischen Universitaet Dresden AöR, Dresden
  - Universitaetsklinikum Duesseldorf AöR, Düsseldorf
  - Goethe University Frankfurt, Frankfurt
  - Universitaetsmedizin Goettingen, Göttingen
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Zentrum Fuer Nieren Hochdruck Und Stoffwechselerkrankungen, Hanover
  - Universitaetsklinikum Heidelberg AöR, Heidelberg
  - Universitaetsklinikum Jena KöR, Jena
  - Universitaetsklinikum Schleswig-Holstein AöR, Kiel
  - Universitaet Leipzig, Leipzig
  - Universitaetsklinikum Schleswig-Holstein AöR, Lübeck
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz KöR, Mainz
  - Klinikum der Technischen Universitaet Muenchen, München
  - LMU Klinikum Muenchen AöR, München
  - Klinikum Der Landeshauptstadt Stuttgart gKAöR, Stuttgart
- Netherlands (3):
  - Universitair Medisch Centrum Groningen, Groningen
  - Leids Universitair Medisch Centrum, Leiden
  - Erasmus Universitair Medisch Centrum Rotterdam, Rotterdam
- Spain (2):
  - Fundacio Hospital Universitari Vall D'Hebron Institut De Recerca, Barcelona
  - Fundacio Puigvert, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muller RU, Guerrot D, Chonchol M, Schmitt R, Uchiyama K, Gansevoort RT, Cornec-Le Gall E. SGLT2 inhibition for patients with ADPKD - closing the evidence gap. Nephrol Dial Transplant. 2025 Nov 26;40(12):2231-2238. doi: 10.1093/ndt/gfaf061. PMID 40199734